CLINICAL TRIAL: NCT02651181
Title: Feasibility Study to Evaluate the Hybrid-Logic Closed Loop System in Type 1 Diabetes -Single-arm, Single-center, in Clinic Study-The DREAMED Trail
Brief Title: Feasibility Study to Evaluate the Hybrid-Logic Closed Loop System in Type 1 Diabetes The DREAMED Trail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC076215ctil
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2017-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Closed Loop System (Experimental)
  Interventions: Device: HLCL- Hybrid Logic Closed Loop System

INTERVENTIONS:
Device: HLCL- Hybrid Logic Closed Loop System — All subjects wearing the HLCL System and using it with the closed loop algorithm

SUMMARY:
Closed loop technology has been shown to reduce both hypoglycemia and hyperglycemia, as well as reduce glycemic variability.

Several groups around the world investigate efforts in developing closed-loop systems. Investigators combined two closed-loop systems with different mode of operation in order to enhance the closed-loop system. The two systems are Hybrid closed-loop system and the MD-Logic closed-loop system . The combined algorithm Hybrid logic closed loop (HLCL) was tested 'In silico' and was proved to be safe and effective. The next step is to test the system in a clinical study in a supervised environment in a camp.

The two systems were tested separately in several clinical studies and were proven to be safe and effective in a diverse population of patients with type 1 diabetes. The MD-Logic system for overnight use "the GlucoSitter" has a CE mark.

The purpose of this study is to collect data on the feasibility of the HLCL system in a camp setting.

DETAILED DESCRIPTION:
Closed loop technology has been shown to reduce both hypoglycemia and hyperglycemia, as well as reduce glycemic variability.

Several groups around the world investigate efforts in developing closed-loop systems. Investigators combined two closed-loop systems with different mode of operation in order to enhance the closed-loop system. The two systems are Hybrid closed-loop system and the MD-Logic closed-loop system . The combined algorithm Hybrid logic closed loop (HLCL) was tested 'In silico' and was proved to be safe and effective. The next step is to test the system in a clinical study in a supervised environment in a camp.

The two systems were tested separately in several clinical studies and were proven to be safe and effective in a diverse population of patients with type 1 diabetes. The MD-Logic system for overnight use "the GlucoSitter" has a CE mark.

The primary objective of the study is to characterize the overall management of the glycemic control using this system including Safety. The data collected in this study will be used to confirm/develop the HLCL System further.

Secondary objectives of this study include evaluation of the HLCL system in a monitored setting (camp) with the following stresses:Exercise, high carbohydrate and high fat meals

This study is a single-arm, single-center, in clinic Investigation in subjects with type 1 diabetes on insulin pump therapy.

Run-in Period:

A total of up to 10 subjects will be enrolled (age 18-40). A minimum of 6 days run-in period with sensor augmented pump will be used to collect sensors and insulin data and to allow the subject to become familiar.

Study Period - Camp:

Following the run-in period subjects will participate in a 5 day, 4 night study period in a camp setting during which the HLCL feature will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes duration > 1 year since diagnosis
* Pump therapy for at least 6 months and Experience with sensor use
* Age 18-40
* A1C <10.0 at time of screening visit
* Willing to follow study instructions
* Willing to perform ≥ 5 finger stick blood glucose measurements daily
* Willing to perform required sensor calibrations
* Patient capable of reading and understand instructions in English

Exclusion Criteria:

* Subject is unable to tolerate tape adhesive in the area of sensor placement
* Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
* Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study drug or device in the last 2 weeks
* Subject has a positive pregnancy screening test
* Subject is female, sexually active without the use of contraception, and plans/able to become pregnant during the course of the study and is not using an acceptable method of contraception
* Subject has had a hypoglycemic seizure within the past 5 months prior to screening visit
* Subject has had hypoglycemia resulting in loss of consciousness within the past 5 months prior to screening visit
* Subject has had an episode of diabetic ketoacidosis within the past 6 months prior to screening visit
* Subject has a history of a seizure disorder
* Subject has central nervous system or cardiac disorder resulting in syncope
* Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
* Subjects with hematocrit lower than the normal reference range or local lab testing
* Subjects with a history or findings on screening electrocardiogram (EKG) of any cardiac arrhythmia, including atrial arrhythmias
* Subjects with a history of adrenal insufficiency
* Subjects with history of migraines that have occurred at least 2 times in the last 3 months prior to enrollment
* Any disease or condition that may influence the A1C testing e.g abnormal red blood cell indices and iron deficiency, sickle cell disease, hemoglobinopathy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Time in range of sensor glucose data between 70 mg/dL to 180 mg/dL, | End of the study- day 5 of the camp
Time in range of sensor glucose data between 70 mg/dL to 180 mg/dL,during night time (12am-6am) | End of the study- day 5 of the camp
Time in range of sensor glucose data between 70 mg/dL to 180 mg/dL,during day time (6am-12am) | End of the study- day 5 of the camp

SECONDARY OUTCOMES:
Event rate of Serious Adverse Events | End of the study- day 5 of the camp
Event rate of Serious Adverse Device Events | End of the study- day 5 of the camp
Event rate of unanticipated Adverse Device Effects | End of the study-day 5 of the camp
Incidence of Diabetic Ketoacidosis | End of the study-day 5 of the camp
Area under the curve of time in the hyperglycemia range | End of the study-day 5 of the camp
Area Under the curve of time in the hypoglycemic range | End of the study-day 5 of the camp
Incidence of Severe Hypoglycemia | End of study -day 5 of the camp

OTHER OUTCOMES:
Percentage of time in Closed Loop | End of study -day 5 of the camp
Total insulin dose | End of study-day 5 of the camp

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, MD, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Medical Center, Petah Tikva, Israel